CLINICAL TRIAL: NCT05813834
Title: US-guided Genicular Nerves Block for Pain Control After Arthroscopic Anterior Cruciate Ligament Repair: A Prospective, Double Blinded, Randomized Controlled Study
Brief Title: Ultrasound-guided Genicular Nerves Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Ismail, Associate Professor of Anesthesia, Surgical ICU and pain management at Faculty of medicine Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-502-2022
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Genicular Nerve Block for Pain in ACL Arthroscopy

STUDY DESIGN:
Intervention Model Description: Genicular Nerves Block
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- genicular nerve block group (Active Comparator): patients will receive genicular nerves block
  Interventions: Procedure: Genicular Nerves Block
- control group (No Intervention): patients will not receive genicular nerves block

INTERVENTIONS:
Procedure: Genicular Nerves Block — US guided genicular nerves block
  Arms: genicular nerve block group

SUMMARY:
Most of arthroscopic ACL repairs are day case surgeries associated with moderate postoperative pain and discomfort. So , finding an effective and safe, analgesic technique with minimal complications is our goal for fast recovery and short hospital stay.

in this study, we aim to compare the efficacy of genicular nerve block against controls on postoperative pain scores, the need for rescue analgesics, patient's satisfaction and range of motion (ROM) after arthroscopic ACL cases.

DETAILED DESCRIPTION:
In this study, we aim to compare the efficacy of genicular nerve block against controls on postoperative pain scores, the need for rescue analgesics, patient's satisfaction and range of motion (ROM) after arthroscopic ACL cases.

ELIGIBILITY:
Inclusion Criteria:

* both genders
* age 18 - 65
* ASA i, ii, iii

Exclusion Criteria:

* ROM less than 90
* advanced renal or liver diseases
* patient refusal
* substance abuse
* site infection
* known sensitivity to any of study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
post operative VAS | 24 hours
  vas score

SECONDARY OUTCOMES:
total morphine consumption | 24 hours
  morphine onsumpton
time to first morphine analgesia | 24 hours
  rescue analgesia
range of motion | 24 hours
  rom
post operative MAP | 24 hours
  map

CONTACTS AND LOCATIONS:
Overall Officials: Dalia K Ismail, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No